CLINICAL TRIAL: NCT01025115
Title: Efficacy of Diamel in the Treatment of Metabolic Syndrome
Brief Title: Diamel in the Treatment of Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Eduardo Cabrera-Rode, National Institute of Endocrinology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-0918-CU
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Metabolic Syndrome
Keywords: Dietary supplement; Diamel; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Diamel
  Interventions: Dietary Supplement: Diamel
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Diamel — Two Diamel tablets (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 12 months, together with the standard treatment for metabolic syndrome consisting in appropriate diet according to patient's weight and physical activity, and appropriate hypertensive drugs (generally ACE inhibitors) for hypertension. Patient´s were also verbally encouraged to increase physical activity (to walk for 30-45 minutes a day 3-4 days a week).
  Arms: A
Dietary Supplement: Placebo — Two Placebo tablets (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 12 months, together with the standard treatment for metabolic syndrome consisting in appropriate diet according to patient's weight and physical activity, and appropriate hypertensive drugs (generally ACE inhibitors) for hypertension. Patient´s were also verbally encouraged to increase physical activity (to walk for 30-45 minutes a day 3-4 days a week).
  Arms: B

SUMMARY:
The purpose of this study is to assess the efficacy of Diamel administration in the treatment of Metabolic Syndrome. The duration of this double-blind placebo controlled phase 3 clinical trial will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome diagnosis according to WHO definition, with or without glucose intolerance.
* Signed informed consent

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes treated with oral hypoglycemic drugs and/or insulin
* Other diseases associated with insulin resistance (eg. Acromegalia, endogenous hypercortisolism, etc)
* Neuropathies or hepatic conditions diagnosed biochemically or by clinical exam.
* Mild or severe heart conditions (eg. heart failure, ischemic cardiopathy)
* Sepsis or any other condition that could potentially interfere with treatment
* Any other treatment that could potentially interfere with treatment
* Pregnancy

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Blood concentrations of glucose at months 0,3,6,9,12. | 12 months
Blood concentrations of insulin at months 0,3,6,9,12. | 12 months
Blood concentrations of cholesterol at months 0,3,6,9,12. | 12 months
Blood concentrations of HDL-cholesterol at months 0,3,6,9,12. | 12 months
Blood concentrations of triglycerides at months 0,3,6,9,12. | 12 months
Blood concentrations of creatinine at months 0,3,6,9,12. | 12 months
Blood concentrations of uric acid at months 0,3,6,9,12. | 12 months

SECONDARY OUTCOMES:
Blood pressure at months 0,3,6,9,12. | 12 months
BMI index at months 0,3,6,9,12. | 12 months
Waist-to-hip index at months 0,3,6,9,12. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cabrera-Rode, PhD, Principal Investigator — National Institute of Endocrinology
Locations (1):
- National Institute of Endocrinology, Havana, La Habana, Cuba